CLINICAL TRIAL: NCT02984839
Title: Incidence of Residual Neuromuscular Blockade in Intra-abdominal Surgery: A Prospective, Observational Study
Status: Completed | Type: Observational
Sponsor: OhioHealth (Other)
Responsible Party: Principal Investigator, Kayla Petersen, Resident Physician, OhioHealth
Other Study IDs: 16-0047
Record Dates: First submitted 2016-12-03; First posted 2016-12-07 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Neuromuscular Blockade; Pulmonary Complication
Keywords: intra-abdominal surgery; neuromuscular blocking agent; post-anesthesia care unit

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intra-abdominal surgery group: The study population will include patients presenting for elective or non-elective intra-abdominal surgery requiring general anesthesia with neuromuscular blockade at OhioHealth Doctors Hospital.
  Quantitative TOF will be recorded by Stimpod NMS450 in PACU.
  Interventions: Device: Stimpod NMS450® Nerve Stimulator, by Xavant™ Technology
- Non-intra-abdominal surgery group: The study population will include patients presenting for elective or non-elective non intra-abdominal surgery requiring general anesthesia with neuromuscular blockade at OhioHealth Doctors Hospital.
  Quantitative TOF will be recorded by Stimpod NMS450 in PACU.
  Interventions: Device: Stimpod NMS450® Nerve Stimulator, by Xavant™ Technology

INTERVENTIONS:
Device: Stimpod NMS450® Nerve Stimulator, by Xavant™ Technology — Quantitative train-of-four (TOF) ratio will be recorded in the post anesthesia care unit (PACU) via Stimpod NMS450

SUMMARY:
The aim of this prospective, observational study is to determine the incidence of post-operative residual neuromuscular blockade (PRNB) in patients undergoing intra-abdominal procedures compared to patients undergoing other noncardiac/non intra-thoracic procedures that also require non-depolarizing neuromuscular blocking agents (NMBA) administration. As intra-abdominal surgeries are independently associated with post-operative pulmonary complications (PPCs), it is important to highlight other factors, such as PRNB, that could contribute to these complications.Although it has been shown that the risk of adverse respiratory events can be reduced by intra-operative quantitative neuromuscular monitoring, such monitoring is not in widespread use.This study will incorporate quantitative monitoring in the post-anesthesia care unit (PACU) setting by using the Stimpod NMS450® in an effort to show a disparity in the incidence of residual paralysis between these two patient populations and to emphasize the need to implement more accurate neuromuscular monitoring, especially for those that are already at increased risk for respiratory complications.

DETAILED DESCRIPTION:
Residual paralysis from non-depolarizing neuromuscular blocking agents (NMBAs) is a common problem that contributes to adverse outcomes in the post-anesthesia care unit (PACU).Unidentified residual neuromuscular blockade (defined as a train-of-four (TOF) ratio <0.9) has been reported in up to 30-42% of patients in the recovery room.Though current literature supports the use of quantitative monitoring of neuromuscular blockade, conventional qualitative TOF count monitoring and clinical signs (head lift, grip strength) continue to be used.There is strong evidence that shows reduction of clinically significant post-operative residual neuromuscular blockade (PRNB) after implementation of quantitative monitoring. Post-operative pulmonary complications (PPCs) are notable adverse outcomes of residual neuromuscular blockade. The implementation of quantitative monitoring may be particularly beneficial to patients who are already predisposed to PPCs secondary to the site of surgery.

The purpose of this study is to evaluate the incidence of PRNB with use of quantitative neuromuscular monitoring in patients undergoing intra-abdominal procedures compared to patients undergoing other surgical procedures that also require NMBA administration.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* ASA physical status classification I-IV
* Procedures requiring intubation and nondepolarizing NMBA administration

  * Laparoscopic surgery
  * Intra-abdominal surgery
  * Procedures using the Da Vinci surgical system
  * Tonsillectomy
  * Septoplasty
  * Shoulder surgery
  * Total hip arthroplasty
  * Carotid endarterectomy
  * Cervical spine surgery
  * Parotidectomy
  * Thyroidectomy
  * Aorto-bifemoral bypass
  * Micro laryngoscopy
  * Nasal or sinus surgery
  * Dental extraction

Exclusion Criteria:

* Non-English speaking population
* ASA V and VI
* Unable to give informed consent
* Cardiac or intra-thoracic procedures performed
* Severe renal insufficiency (Serum Creatinine >2.0 mg/dL)
* Severe hepatic dysfunction
* Underlying neuromuscular disease
* Currently enrolled in another therapeutic study
* Pregnant patients at any stage of pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include all patients age 18 or older with American Society of Anesthesiologists (ASA) physical status I-IV presenting for elective or non-elective surgery requiring general anesthesia with neuromuscular blockade.While previous studies have found that up to 30-42% of patients experience PRNB in the PACU, no previous studies have estimated the incidence of PRNB by surgical procedure (i.e., intra-abdominal versus other surgical procedures).Therefore, this study will be more descriptive in nature.A difference of at least 10% in the incidence of PRNB between the two groups will be considered clinically significant.A maximum number of 120 (approximately 60 patients who undergo intra-abdominal surgery and 60 patients who undergo non intra-abdominal surgical procedures) will be enrolled during the course of the study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-11; Primary Completion 2017-03-21 (Actual); Study Completion 2017-05-16 (Actual)

PRIMARY OUTCOMES:
Train-of-four (TOF) ratio | 15 minutes post arrival in the post anesthesia care unit (PACU)
  Average TOF ratio will be calculated from two consecutive readings using the Stimpod NMS450 within 15 minutes of arrival in the PACU

SECONDARY OUTCOMES:
Need for supplemental O2 therapy | 30 minutes post arrival in the PACU
  Necessity for supplemental O2 therapy after 30 minutes in PACU will be recorded via chart review to determine post operative pulmonary complication

CONTACTS AND LOCATIONS:
Overall Officials: Kayla Petersen, D.O., Principal Investigator — Resident Physician
Locations (1):
- OhioHealth Doctors Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No